CLINICAL TRIAL: NCT05714098
Title: Gerofit Exercise Intervention for Older Adults With Sickle Cell Disease (SICKLE-FIT Study)
Acronym: SICKLE-FIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00111833
Record Dates: First submitted 2023-01-18; First posted 2023-02-06 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell anemia; older adults; exercise; geriatrics; functional impairment
MeSH Terms: conditions — Anemia, Sickle Cell; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): Each cohort of 5-8 participants will exercise 3 days a week for up to 12 weeks. Exercise sessions will be virtual
  Interventions: Behavioral: Gerofit Exercise Program

INTERVENTIONS:
Behavioral: Gerofit Exercise Program — The tele-Gerofit exercise intervention has training focused on meeting the physical activity guidelines and incorporating cardiovascular, strength, and balance training. Sessions will also include a mindfulness component, warm up, cool-down, and safety checks. Exercises are personalized to each person's functional status. Intensity of exercises will be determined by participants providing a rating of perceived exertion (RPE) on a scale of 0 (easy) to 10 (very hard) throughout the session. Initial exercise sessions will start at low-intensity and will gradually increase the duration and intensity to allow each person to reach recommended exercise levels at their own pace. Exercises are done virtually via Zoom. Each cohort will have 5-8 participants. The exercise program will be optimized after each cohort with modifications based on participant and exercise expert feedback.

SUMMARY:
The purpose of this study to assess the feasibility, acceptability, and safety of a personalized exercise training program adapted from Gerofit to improve physical health and quality of life for adults with SCD

DETAILED DESCRIPTION:
The purpose of this study is to adapt and pilot the Gerofit personalized exercise intervention for older adults with sickle cell disease (age ≥ 40 years). The Sickle Cell Disease Functional Assessment (SCD-FA) will be performed at steady state at baseline and every 3 months to track progress. Endpoints include feasibility, acceptability, and safety. All participants will be interviewed to identify barriers and facilitators to exercise and how to better optimize the exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of sickle cell disease (any genotype) confirmed by hemoglobin electrophoresis, high performance liquid chromatography, or genotyping
* Understand and speak fluent English.

Exclusion Criteria:

* Diagnosed with moderate or severe cognitive impairment based on ICD-10 codes or report from their outpatient provider
* Unable to self-consent
* Wheelchair-bound
* Successfully treated with hematopoietic stem cell transplantation for SCD
* Have moderate to severe uncorrected visual or auditory impairment
* Oxygen-dependent
* Pregnant
* Have severe avascular necrosis requiring an assist device
* Unstable cardiac disease.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-08-08 (Actual)

PRIMARY OUTCOMES:
Feasibility, as measured by number of participants completing at least 50% of the exercise sessions | 12 weeks

SECONDARY OUTCOMES:
Safety, as measured by number of participants with moderate or severe adverse events | 12 weeks
  Number of participants with 1 or more moderate or severe adverse events within 48 hours after each exercise session
Acceptability, as measured by acceptability survey | 12 weeks
  Number of participants reporting the intervention as acceptable

OTHER OUTCOMES:
Change in mobility as measured by Usual Gait Speed | Baseline, 12 weeks, 24 weeks
Change in balance as measured by Timed Up and Go | Baseline, 12 weeks, 24 weeks
Change in aerobic endurance as measured by Six-Minute Walk Test | Baseline, 12 weeks, 24 weeks
Change in upper body strength as measured by grip strength | Baseline, 12 weeks, 24 weeks
Change in lower body strength as measured by 30-second chair stand | Baseline, 12 weeks, 24 weeks
Change in quality of movement measured by functional movement screen | Baseline, 12 weeks. 24 weeeks

CONTACTS AND LOCATIONS:
Overall Officials: Charity I Oyedeji, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morey MC, Lee CC, Castle S, Valencia WM, Katzel L, Giffuni J, Kopp T, Cammarata H, McDonald M, Oursler KA, Wamsley T, Jain C, Bettger JP, Pearson M, Manning KM, Intrator O, Veazie P, Sloane R, Li J, Parker DC. Should Structured Exercise Be Promoted As a Model of Care? Dissemination of the Department of Veterans Affairs Gerofit Program. J Am Geriatr Soc. 2018 May;66(5):1009-1016. doi: 10.1111/jgs.15276. Epub 2018 Feb 12. PMID 29430642
- [Background] Oyedeji CI, Hall K, Luciano A, Morey MC, Strouse JJ. The Sickle Cell Disease Functional Assessment (SCD-FA) tool: a feasibility pilot study. Pilot Feasibility Stud. 2022 Mar 4;8(1):53. doi: 10.1186/s40814-022-01005-3. PMID 35246265
- [Background] Morey MC, Pieper CF, Crowley GM, Sullivan RJ, Puglisi CM. Exercise adherence and 10-year mortality in chronically ill older adults. J Am Geriatr Soc. 2002 Dec;50(12):1929-33. doi: 10.1046/j.1532-5415.2002.50602.x. PMID 12473002
- [Background] Morey MC, Cowper PA, Feussner JR, DiPasquale RC, Crowley GM, Kitzman DW, Sullivan RJ Jr. Evaluation of a supervised exercise program in a geriatric population. J Am Geriatr Soc. 1989 Apr;37(4):348-54. doi: 10.1111/j.1532-5415.1989.tb05503.x. PMID 2921457
- [Background] Oyedeji C, Strouse JJ, Crawford RD, Garrett ME, Ashley-Koch AE, Telen MJ. A multi-institutional comparison of younger and older adults with sickle cell disease. Am J Hematol. 2019 Apr;94(4):E115-E117. doi: 10.1002/ajh.25405. Epub 2019 Jan 31. No abstract available. PMID 30663090
- [Background] Liem RI. Balancing exercise risk and benefits: lessons learned from sickle cell trait and sickle cell anemia. Hematology Am Soc Hematol Educ Program. 2018 Nov 30;2018(1):418-425. doi: 10.1182/asheducation-2018.1.418. PMID 30504341
- [Background] Merlet AN, Messonnier LA, Coudy-Gandilhon C, Bechet D, Gellen B, Rupp T, Galacteros F, Bartolucci P, Feasson L. Beneficial effects of endurance exercise training on skeletal muscle microvasculature in sickle cell disease patients. Blood. 2019 Dec 19;134(25):2233-2241. doi: 10.1182/blood.2019001055. PMID 31742587
- [Background] Liem RI, Akinosun M, Muntz DS, Thompson AA. Feasibility and safety of home exercise training in children with sickle cell anemia. Pediatr Blood Cancer. 2017 Dec;64(12). doi: 10.1002/pbc.26671. Epub 2017 Jun 9. PMID 28598539

DOCUMENTS (1):
  • Informed Consent Form (2025-01-09): https://cdn.clinicaltrials.gov/large-docs/98/NCT05714098/ICF_000.pdf